CLINICAL TRIAL: NCT00839059
Title: Open-Label, Multi-Center Phase I Dose-Escalation Study With Lenalidomide In Patients With Acute Myeloid Leukemia
Brief Title: Lenalidomide In Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Results of an interim analysis and a hardly ongoing enrolment in the last 10 months in all six participating centres
Sponsor: University of Ulm (Other)
Responsible Party: Prof. Dr. Reinhard Marre, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG08-07
Record Dates: First submitted 2009-01-20; First posted 2009-02-09 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; lenalidomide
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Dose escalation:
  Level 0 to level 5, starting with level 1 = 25mg lenalidomide per os daily, Cohorts of 3 patients (to be expanded up to 6 if 1 DLT is observed among the first 3 patients) will be sequentially allotted to progressively higher dose levels of lenalidomide on the basis of the presence and severity of lenalidomide related toxicity encountered in the first cycle or lenalidomide related serious adverse reactions.
  Duration of the first cycle: 56days, each following cycle will last 28 days

SUMMARY:
This is a Phase I, open-label, multi-center, dose-escalation study of lenalidomide in adult patients with newly diagnosed, relapsed or refractory acute myeloid leukemia. All patients will receive lenalidomide per oral daily (starting dose is 25 mg/d). Cohorts of 3 patients (to be expanded up to 6 if 1 dose-limiting toxicity (DLT) is observed among the first 3 patients) will be sequentially allotted to progressively higher dose levels of lenalidomide on the basis of the presence and severity of lenalidomide-related toxicity or lenalidomide related serious adverse reactions encountered in the first cycle. For the purpose of this study, patients' enrollment will continue until the maximum tolerated dose (MTD) will be determined and characterized.

ELIGIBILITY:
Inclusion Criteria:

Disease state:

* Age > 70 years newly diagnosed AML (including de novo, s-AML, t-AML)considered ineligible for intensive treatment. Ineligibility for intensive treatment has to be documented within the case report forms (Medical/Oncologic History).
* Age > 60 years relapsed/refractory AML in medically fit patients and newly diagnosed AML (including de novo, s- AML,t-AML) in medically unfit patients
* Age 18-60 years: second or higher relapse of AML, not eligible for intensive therapy
* WBC <20x109/l, pretreatment with hydroxyurea is allowed to lower WBC
* Prior chemo-immunotherapy and other study-medications must have been completed 2 weeks before study treatment start. Treatment with hydroxyureas should be discontinued 1 day before initiating dosing with lenalidomide
* Willingness and ability to comply with scheduled visits,treatment plan, laboratory tests and other study procedures
* Females of childbearing potential (FCBP)† must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from - FCBP must have two negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting study drug.
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Acute promyelocytic leukemia [t(15;17)]
* bleeding disorder independent of the AML
* uncontrolled infection
* insufficiency of the kidneys (creatinin >1.5x upper normal serum level), of the liver (bilirubin, AST or AP > 2x upper normal serum level)
* severe obstructive or restrictive ventilation disorder
* heart failure NYHA III/IV
* severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* no consent for registration, storage and processing of the individual disease-characteristics and course
* peripheral neuropathy
* Performance status WHO > 2
* Presence of any medical/psychiatric condition or laboratory abnormalities which may limit full compliance with the study, increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study
* Pregnancy or breast-feeding
* Known positive for HIV or infectious hepatitis, type A, B or C
* Known hypersensitivity to thalidomide
* Any prior use of lenalidomide
* Drug or alcohol abuse within the last 6 months
* Participating in other studies within the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLTs), Maximum tolerated dose (MTD) | 1-56 days

SECONDARY OUTCOMES:
Measurement of the pharmacokinetic profile of lenalidomide | 1st and 8th day
Objective tumor response, as defined using the revised recommendations of the International Working Group for diagnosis, standardization of response criteria in Acute Myeloid Leukemia for AML | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schlenk, MD, Principal Investigator — University Hospital of Ulm
Locations (6):
- Germany (6):
  - University Hospital of Bonn, Bonn
  - University Hospital of Düsseldorf, Düsseldorf
  - Hospital of the Johann Wolfgang Goethe University, Frankfurt
  - University Hospital of Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University Hospital of Ulm, Ulm

REFERENCES:
- See also: Related Info — http://www.kompetenznetz-leukaemie.de